CLINICAL TRIAL: NCT03792854
Title: Prospective Observational Trial to Evaluate Quality of Life After Definitive Chemoradiation in Patients With Anal Cancer (LANACARE)
Acronym: LANACARE
Status: Recruiting | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Falk Roeder, Consultant, Ludwig-Maximilians - University of Munich
Other Study IDs: V1 10/2018
Record Dates: First submitted 2019-01-02; First posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Anal Cancer; Quality of Life; Chemoradiation
Keywords: anal cancer; quality of life; chemoradiation
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: EORTC QLQ C30 — standardized questionaire
Other: EORTC QLQ CR29 — standardized questionaire

SUMMARY:
Observational study to evaluate longitudinal quality of life according to standardized EORTC questionaires as well as functional outcome, oncological outcome and toxicity in patients treated with definitive chemoradiation for anal cancer

DETAILED DESCRIPTION:
Observational study to evaluate longitudinal quality of life according to standardized EORTC questionaires as well as functional outcome, oncological outcome and toxicity in patients treated with definitive chemoradiation for anal cancer. Qol will be evaluated by standardized EORTC questionaires QLQ C30 and QLQ CR29. Acute and late toxicity will be assessed according to CTCAE 4.03. Oncological outcome will be assessed with regard to local and distant control, patterns of recurrence, freedom from treatment failure and overall survival. Correlations of physicians- and patients-assessed functional outcomes are planned.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven anal cancer without distant metastases
* indication for definitive chemoradiation therapy based on multidisciplinary evaluation
* age >=18 years
* written informed consent
* ability to answer the standardized questionaires according to the treating physician

Exclusion Criteria:

* age < 18 years
* prior systemic therapy with regard to anal cancer
* distant metastases
* second malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: see eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Qol (EORTC QLQC30) absolute values and change over time | day 0, end of week 6, 12, 19, 32, 58, 84, 110, 162, 214, 266
  Quality of life measured by EORTC questionaire QLQC30 in absolute values at different time points and change over time
Qol (EORTC QLQCR29) absolute values and change over time | day 0, end of week 6, 12, 19, 32, 58, 84, 110, 162, 214, 266
  Quality of life measured by EORTC questionaire QLQCR29 in absolute values at different time points and change over time

SECONDARY OUTCOMES:
local control | end of week 6, 12, 19, 32, 58, 84, 110, 162, 214, 266
  absence of disease progression inside the target volume of radiation therapy
distant control | end of week 6, 12, 19, 32, 58, 84, 110, 162, 214, 266
  absence of disease progression outside the target volume of radiation therapy
freedom from treatment failure | end of week 6, 12, 19, 32, 58, 84, 110, 162, 214, 266
  absence of disease progression inside or outside the target volume of radiation therapy
overall survival | end of week 6, 12, 19, 32, 58, 84, 110, 162, 214, 266
  absence of death from any cause
acute toxicity | day 0, end of week 6, 12, 19
  acute toxicity caused by chemoradiation according to CTCAE 4.03
late toxicity | end of week 32, 58, 84, 110, 162, 214, 266
  late toxicity caused by chemoradiation according to CTCAE 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Falk Roeder, MD, Principal Investigator — Ludwig-Maximilians Universität München
Locations (1):
- Department of Radiation Oncology, University Hospital, LMU Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No